CLINICAL TRIAL: NCT06363084
Title: Nimotuzumab Plus Adjuvant Chemotherapy vs Adjuvant Chemotherapy Alone for Resectable Pancreatic Cancer: a Propensity Score Matching Analysis
Brief Title: A Retrospective Study for Nimotuzumab Plus Postoperative Adjuvant Chemotherapy for Resectable Pancreatic Cancer
Status: Completed | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IST-Nim-PC-6
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-03

CONDITIONS: Resectable Pancreatic Cancer
MeSH Terms: interventions — nimotuzumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study arm: Nimotuzumab plus adjuvant chemotherapy
  Interventions: Drug: Nimotuzumab
- control arm: adjuvant chemotherapy alone (without Nimotuzumab)

INTERVENTIONS:
Drug: Nimotuzumab — Nimotuzumab (400mg) was given weekly
  Other Names: Taixinsheng
  Groups: study arm

SUMMARY:
This trial is a retrospective, observational study, patients who underwent surgical resection of the pancreas for non-metastatic pancreatic cancer between 2016 and 2022 were selected and divided into two groups according to with (study arm) or without (control arm) nimotuzumab. The primary efficacy endpoint was overall survival (OS).

DETAILED DESCRIPTION:
This trial is a retrospective, observational study based on real-world data obtained from the Health Information System (HIS) of Ruijin Hospital, Shanghai Jiao Tong University School of Medicine. Patients who underwent surgical resection of the pancreas for non-metastatic pancreatic cancer between 2016 and 2022 were selected and divided into two groups according to with (study arm) or without (control arm) nimotuzumab. The primary efficacy endpoint was overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years old, gender is not limited;
* Confirmed by histopathological or cytological diagnosis of pancreatic cancer;
* Underwent surgical resection of the pancreas for non-metastatic pancreatic cancer (including resectable/borderline resectable pancreatic cancer, or locally advanced pancreatic cancer);
* Received Nimotuzumab plus adjuvant chemotherapy or adjuvant chemotherapy alone after surgery.

Exclusion Criteria:

* Patients with other primary malignancies other than pancreatic cancer;
* Evidence of recurrence or distant metastasis before surgery
* Received immunotherapy drugs (such as PD-1 inhibitors, etc.) used during adjuvant therapy, or proprietary Chinese medicines with anti-tumor indications, or hyperthermia, targeted therapy drugs other than nimotuzumab;
* Key information is missing (e.g., primary endpoint data were not available).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who underwent surgical resection of the pancreas for non-metastatic pancreatic cancer
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
overall survival (OS） | approximately 84 months
  The primary endpoint is overall survival (OS), defined as the time from the start of surgery to the date of death due to any cause.

SECONDARY OUTCOMES:
disease-free survival (DFS) | approximately 84 months
  DFS is defined as the time from surgical resection to the first tumor recurrence/progression or death due to any cause.
locoregional recurrence-free survival (LRRFS) | approximately 84 months
  LRRFS is defined as the time from surgical treatment to clinically or radiographically confirmed local recurrence and/or regional progression at follow-up.

IPD SHARING:
Plan to Share IPD: No